CLINICAL TRIAL: NCT05146635
Title: Optimal Adjuvant Intravesical Therapy for Intermediate Risk Non Muscle Invasive Bladder Cancer: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Lecturer of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AE-12-2021
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Intravesical therapy; Recurrence; Progression
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence; Disease Progression | interventions — Epirubicin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravesical immunotherapy (BCG) group (Active Comparator)
  Interventions: Drug: Intravesical Bcg
- Intravesical chemotherapy (Epirubicin) group (Active Comparator)
  Interventions: Drug: Intravesical chemotherapy (epirubicin)

INTERVENTIONS:
Drug: Intravesical Bcg — Patients will receive induction and maintenance BCG after complete TURBT.
  Arms: Intravesical immunotherapy (BCG) group
Drug: Intravesical chemotherapy (epirubicin) — Patients will receive induction and maintenance epirubicin after complete TURBT.
  Arms: Intravesical chemotherapy (Epirubicin) group

SUMMARY:
The objective of this prospective, single-center randomized controlled trial is to identify the optimal adjuvant intravesical therapy in patients with intermediate risk (IR) non muscle invasive bladder cancer by comparing two commonly utilized intravesical regimens; intravesical immunotherapy (BCG) and intravesical chemotherapy.

DETAILED DESCRIPTION:
Bladder cancer (BC) represents a frequent urologic malignancy, and is mainly diagnosed as non-muscle invasive, At presentation, approximately 30% of patients have muscle-invasive BC (clinical T2 or higher) .

Both the natural history of non-muscle-invasive bladder cancer (NMIBC) and its treatment strategies are highly variable. Although some patients never experience disease recurrence, others experience disease progression and eventually die of their disease .

In the absence of intravesical treatment, a patient with non-muscle-invasive BC has a 47% probability of disease recurrence within 5 years of diagnosis and a 9% probability of progression to muscle-invasive disease .

Low-, intermediate- and high-risk categories have been defined to help guide the treatment of patients with NMIBC (Ta, T1, and CIS). Treatment of NMIBC is now relatively well-defined for high-risk and low-risk disease presentation, and awaits further refinement through improvements in therapeutic options .

Solitary low-grade tumors, especially smaller lesions (3 cm or less), respond best to resection and immediate instillation of intravesical agents, whereas higher risk lesions, such as carcinoma in situ and high-grade T1 stage disease, have demonstrated good response to BCG when given on a schedule of induction (an initial 6-week course) and maintenance (3-weekly courses every 6 months for 3 years) .

However, while low- and high-risk diseases have been well-classified, the intermediate-risk (IR) category has traditionally comprised a heterogeneous group of patients that do not fit into either of these categories . As a result, many urologists remain uncertain about the categorization of patients as 'intermediate-risk' as well as the selection of the most appropriate therapeutic option for this patient population .

The pathology of IR NMIBC has been defined by different organizations (American Urological Association, European Association of Urology, National Comprehensive Cancer Network, and International Consultation on Urological Diseases) as those patients with recurrent (<1 year) low-grade Ta disease, solitary low-grade Ta >3cm, multifocal low-grade Ta disease or high-grade Ta disease <3 cm .

Current recommendations for therapy from the aforementioned organizations suggest a basic role for induction and maintenance therapy with either immunotherapy or chemotherapy. Data from a number of recent trials suggest that BCG with maintenance is superior to maintenance chemotherapy in this population as regard to recurrence free survival. On the other hand, no significant benefit of BCG compared with chemotherapy for tumor progression was identified.

Most of these studies were limited by its heterogeneity of patients (non-standardized definition of IR) and non-unified regimen of intravesical treatment (course or utilized chemotherapeutic agent). A well-designed randomized controlled trial with a rigorous methodology is warranted to provide a solid evidence for best practice in this special group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged >18 years)
* Patients with primary or recurrent papillary NMIBC.
* Complete TURBT.
* Patients with IR NMIBC confirmed by histopathology.

Exclusion Criteria:

* Inability to give informed consent.
* Patients with history of previous radiotherapy or systemic chemotherapy.
* Patients suffering from immuno-deficiency or other malignancies.
* Patients with history of hypersensitivity reaction to BCG or epirubicin.
* Examination under anesthesia (EUA) reveals palpable bladder mass.
* Patients with low or high risk NMIBC by histopathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence rate | 2 years
  Number of patient who will develop Recurrence rate during follow up
Tumor Progression rate | 2 years
  Number of patient who will develop Progression rate during follow up

SECONDARY OUTCOMES:
Side effects from intravesical treatments | 2 years
  Side effects from intravesical treatments

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Mansoura University
Locations (1):
- Mansoura Urology and Nephrology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided